CLINICAL TRIAL: NCT06826612
Title: A Phase 1/2, Randomized, Sequential, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Efficacy of a One-Time, Bilateral, Intraparenchymal Infusion of SPK-10001 Into the Caudate and Putamen in Participants With Huntington's Disease
Brief Title: A Randomized Study of SPK-10001 Gene Therapy in Participants With Huntington's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPK-10001-101
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-07

CONDITIONS: Huntington Disease
Keywords: Huntington's Disease; SPK-10001; Adult-onset HD; HD; Rare Disease; Chorea; Movement Disorder; Spark Therapeutics; Cognition; Gene Therapy; AAV; mHTT
MeSH Terms: conditions — Huntington Disease; Rare Diseases; Chorea; Movement Disorders

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 4 sequential parts.
  * Part A is an open-label cohort in which all participants will receive SPK-10001.
  * Part B is randomized, double-blind and placebo-surgery-controlled.
  * Part C is a crossover open-label portion where participants who received placebo-surgery control in Part B will receive SPK-10001.
  * Part D is long term follow-up after completion of active treatment in any of Parts A, B, or C.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Part A is open-label and non-randomized.
  * Part B is blinded and randomized.
  * Part C is open-label and non-randomized.
  * Part D is open-label and non-randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SPK-10001 (Experimental)
  Interventions: Genetic: SPK-10001
- Placebo Surgery Control (Other)
  Interventions: Other: Placebo Surgery Control

INTERVENTIONS:
Genetic: SPK-10001 — Specified dose on specified days
  Arms: SPK-10001
Other: Placebo Surgery Control — Placebo Surgery procedure for SPK-10001
  Arms: Placebo Surgery Control

SUMMARY:
The main goal of this study is to evaluate the safety, tolerability, and preliminary efficacy of SPK-10001 in participants with Huntington's Disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Have confirmed huntingtin (HTT) cytosine-adenine-guanine (CAG) repeat length ≥40 on genetic testing and confirmation diagnostic test by the central laboratory (CL) at screening.
* Have striatal atrophy demonstrated by caudate/intracranial volume less than the age-adjusted cutoff values associated with HDISS Stage 1.
* Have UHDRS Total Motor Score (TMS) equal to or greater than the age-adjusted cutoff value associated with HDISS Stage 2.
* Have UHDRS Total Functional Capacity (TFC) greater than or equal to 11.
* Use of cholinesterase inhibitors, memantine, amantadine, or riluzole must have been at stable dosing for at least 12 weeks before screening and baseline and anticipated to remain stable during the first 12 months after SPK-10001 administration.
* Antidepressant or benzodiazepine use must have been at stable dosing for at least 12 weeks before screening and baseline and anticipated to remain stable during the first 12 months after SPK-10001 administration.
* Antipsychotics for motor symptoms or mood stabilization (i.e., irritability or aggressive behavior) and/or tetrabenazine, valbenazine, or deutetrabenazine must have been at a stable dose for at least 12 weeks before screening and baseline and are anticipated to remain stable during the first 12 months after SPK-10001 administration.

Key Exclusion Criteria:

* A safe trajectory is not able to be identified for targeting placement of the cannula into the caudate or putamen on both sides of the brain due to extent of atrophy or other anatomical features.
* Have received an antisense oligonucleotide therapy during the past year.
* History of deep brain stimulation.
* History of or intention to undergo gene therapy, cell transplantation, or brain surgery during the course of the study.
* Have participated in an investigational drug study with a systemic administration within 6 weeks or 5 half-lives of screening, whichever is longer.

Additional protocol-defined inclusion/exclusion criteria apply.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2035-01-12 (Estimated); Study Completion 2035-01-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 up to approximately 5 years
Severity of TEAEs | Day 1 up to approximately 5 years
Change from Baseline in Unified Huntington's Disease Rating Scale (UHDRS®) Total Functional Capacity (TFC) Score | Baseline, Month 24

SECONDARY OUTCOMES:
Change from Baseline in Motor Symptom Progression Based on Huntington's Disease Digital Motor Score (HDDMS) | Baseline, Months 12, 18, and 24
Change from Baseline in Composite UHDRS (cUHDRS) Score | Baseline, Months 12, 18, and 24
Change from Baseline in UHDRS TFC Score | Baseline, Months 12 and 18

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Cincinnati/Cincinnati Children's Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburg, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No